CLINICAL TRIAL: NCT01496612
Title: A Phase Two Clinical Trial of Buspirone Therapy in Localization-Related Epilepsy
Brief Title: Buspirone Therapy for Localized Epilepsy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 120033; 12-N-0033
Record Dates: First submitted 2011-12-17; First posted 2011-12-21 (Estimated); Results first posted 2021-09-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2016-04-19

CONDITIONS: Anxiety Disorder; Seizures; Epilepsy; Partial Epilepsy; Depression
Keywords: Epilepsy; Temporal Lobe Epilepsy; Serotonin 1A Receptor; Seizures
MeSH Terms: conditions — Anxiety Disorders; Seizures; Epilepsy; Epilepsies, Partial; Depression; Epilepsy, Temporal Lobe | interventions — Buspirone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Phase (Experimental)
  Interventions: Drug: Buspirone
- Alternate Study Phase (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buspirone
  Arms: Study Phase
Drug: Placebo
  Arms: Alternate Study Phase

SUMMARY:
Background:

Buspirone is a drug that is approved for the treatment of anxiety in adults. Studies suggest that buspirone might act on parts of the brain that can increase certain levels of brain activity. Increasing this brain activity may help decrease epileptic seizures that come from certain parts of the brain. Researchers want to see if buspirone can reduce seizure frequency in people with seizures who are already taking antiseizure medication.

Objectives:

To test whether buspirone can reduce the frequency of seizures in people whose seizures seem to start from one part of the brain.

Eligibility:

Individuals between 18 and 65 years of age who have seizures coming from one or more places in the brain.

Participants must have tried at least two different antiseizure medications.

Participants must also have had at least three seizures during a 1-month observation period while on current medicines.

Design:

Participants will have a screening visit with a physical exam and medical history. Participants will complete mood and memory testing scales. Blood, urine, and saliva samples will be collected.

Participants will have a magnetic resonance imaging scan to evaluate brain structures that relate to epilepsy. They will also have a positron emission tomography scan to look at parts of the brain that are affected by buspirone.

Participants will start taking a study drug (either buspirone or placebo) twice daily. They will keep a calendar of seizures and record any side effects. Treatment will be monitored with clinic visits and blood samples.

After 12 weeks on the study drug, participants will gradually stop taking either the placebo or buspirone over two weeks. They will stay off the drug for another 2 weeks.

After 2 weeks, participants will start taking a study drug that is the opposite of the one they had before. They will keep a calendar of seizures and record any side effects. Treatment will be monitored with clinic visits and blood samples.

After 12 weeks on the study drug, participants will gradually stop taking either the placebo or buspirone.

Participants will have a final followup visit with additional blood tests, mood and memory testing scales and imaging studies.

DETAILED DESCRIPTION:
OBJECTIVE:

To initiate a pilot clinical trial assessing the safety, tolerability and efficacy of the 5HT1A receptor agonist buspirone in patients with localization-related epilepsy. Buspirone is a 5HT1A receptor agonist that is approved for the treatment of anxiety disorders. Patients with localization-related epilepsy have reduced 5HT1A receptor binding on 18FCWAY positron emission tomography (PET). Increasing neurotransmitter activity at 5HT1A receptor sites may ameliorate seizures.

STUDY POPULATION:

Forty patients with localization-related epilepsy

DESIGN:

A randomised, double-blind, placebo-controlled cross-over, phase II clinical trial.

The trial will have a screening phase in which each patient will undergo physical and neurological examination, and standard blood tests, followed by a one month baseline phase. At the end of baseline, patients who qualify will have neuropsychological, anxiety, and mood evaluation, FCWAY PET and MRI (if imaging was not performed already). During the subsequent first study phase, patients will be randomized to buspirone or matching placebo. After completion of the first study phase, patients will be crossed over to the alternate study arm. At the end of the study, any patient who wishes to do so may remain on open-label buspirone.

OUTCOME MEASURES:

1. Difference in seizure rate comparing the 3 month placebo and active study phases
2. Neuropsychological, anxiety, and mood indices comparing the 3 month placebo and active study drug phases

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients may be male or female.
* Patients will be aged 18 65
* Patients must have at least 3 seizures during the one-month baseline.
* Localization-related epilepsy diagnosed by standard clinical criteria that has not responded to treatment with two standard antiepileptic drugs either sequentially or in combination.
* Patients must be able to provide informed consent
* Patients must be able to remain on their baseline AED drugs and doses throughout the study
* Patients must be able to use seizure calendars to record seizures throughout the trial.

EXCLUSION CRITERIA:

* Pregnant patients will not participate in the study.
* During the study, women of child-bearing potential must use a reliable method of birth control and will have pregnancy testing throughout the protocol.
* Use of any alcohol or recreational drugs starting two weeks before entering baseline and for the duration of the study.
* Patients on medications with potential for a clinically significant interaction with buspirone, including MAO inhibitors, clozapine, zolpidem, hypnotics, hydromorphone derivatives, oxycodone, and diltiazem.
* Current treatment for psychiatric disorder other than depression, anxiety or bipolar disorder.
* Patients with a diagnosis of schizophrenia.
* Current treatment for another significant medical disorder, such as diabetes, or heart disease, or an untreated disorder, that might interfere with the study.
* Calculated Creatinine clearance of less than 80 ml/min calculated with the Cockcroft-Gault formula:
* Clcr = [(140-age) times ideal body weight in Kg] times (0.85 if female) divided by (72 times serum Cr in mg/dL)
* Evidence of impaired liver function based on serum chemistries.
* Inability to participate in the study procedures, such as MRI, PET, seizure and adverse event recording, or drug titration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-11-22; Primary Completion 2016-04-19 (Actual); Study Completion 2016-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William H Theodore, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Alper K, Schwartz KA, Kolts RL, Khan A. Seizure incidence in psychopharmacological clinical trials: an analysis of Food and Drug Administration (FDA) summary basis of approval reports. Biol Psychiatry. 2007 Aug 15;62(4):345-54. doi: 10.1016/j.biopsych.2006.09.023. Epub 2007 Jan 16. PMID 17223086
- [Background] Berg AT, Berkovic SF, Brodie MJ, Buchhalter J, Cross JH, van Emde Boas W, Engel J, French J, Glauser TA, Mathern GW, Moshe SL, Nordli D, Plouin P, Scheffer IE. Revised terminology and concepts for organization of seizures and epilepsies: report of the ILAE Commission on Classification and Terminology, 2005-2009. Epilepsia. 2010 Apr;51(4):676-85. doi: 10.1111/j.1528-1167.2010.02522.x. Epub 2010 Feb 26. PMID 20196795
- [Background] Bhagwagar Z, Rabiner EA, Sargent PA, Grasby PM, Cowen PJ. Persistent reduction in brain serotonin1A receptor binding in recovered depressed men measured by positron emission tomography with [11C]WAY-100635. Mol Psychiatry. 2004 Apr;9(4):386-92. doi: 10.1038/sj.mp.4001401. PMID 15042104

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from referrals to the NINDS Clinical Epilepsy Section. In addition, self-referral was permitted.
Pre-assignment Details: Nine participants were consented to the protocol. Two participants decided not to participate prior to baseline and randomization.
Groups:
- Buspirone Then Placebo: Participants were administered Buspirone, followed by a washout period, and then administered Placebo
- Placebo Then Buspirone: Participants were administered Placebo, followed by a washout period, and then administered Buspirone
Period: 1st Intervention
Arm/Group | Buspirone Then Placebo | Placebo Then Buspirone
Started | 3 | 4
Completed | 1 | 4
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: 2nd Intervention
Arm/Group | Buspirone Then Placebo | Placebo Then Buspirone
Started | 1 | 4
Completed | 1 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants enrolled in the study
Arm/Group | All Participants
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Seizure Frequency in the Buspirone (Active) and Placebo Periods
Description: Participants utilized a seizure calendar to record the number of seizures that occurred during the three month treatment period, i.e., while participants were either taking Buspirone or Placebo. Seizure frequency was calculated as the total number of seizures occurring during each three month period. For each period a mean was calculated across subjects.
Time Frame: Three months
Measure: Mean (Standard Deviation); unit: number of seizures
Groups:
- Buspirone: Participants with epilepsy receiving Buspirone
- Placebo: Participants with epilepsy receiving Placebo
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 5 | 5
number of seizures | 33.2 (25.51) | 31.2 (32.57)

2. Secondary Outcome: Mean Score on the Hamilton Anxiety Rating Scale (HAM-A) at the End of the Active and Placebo Periods.
Description: Participants were administered the Hamilton Anxiety Rating Scale (HAM-A) at the end of each three month treatment period, i.e., while participants were either on Buspirone or Placebo. The HAM-A measures an individual's severity of anxiety symptoms. The scale consists of 14 parameters, each deﬁned by a series of symptoms. Each group of symptoms is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild anxiety, 18-24 mild to moderate anxiety and 25-30 moderate to severe anxiety.
Time Frame: Three months
Population: One participant in the Placebo group did not complete the HAM-A scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 5 | 4
score on a scale | .80 (.45) | 2 (.82)

3. Secondary Outcome: Mean Score on the Hamilton Depression Rating Scale (HAM-D) at the End of the Active and Placebo Periods
Description: The Hamilton Depression Rating Scale (HAM-D) was administered to participants at the end of each treatment period. The HAM-D is a multiple item questionnaire used to provide an indication of depression. The questionnaire is designed for adults and is used to rate the severity of their depression by probing mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms. Although the HAM-D form lists 21 items, the scoring is based on the ﬁrst 17 items. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine items are scored from 0-2 with 0 = absent and 2 = frequent or severe. Scores range from 0 to 50 with a score of 0-7 representing normal and a score >/= 23 representing very severe depression.
Time Frame: Three months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 5 | 5
score on a scale | 1.40 (1.14) | 2.40 (1.82)

4. Secondary Outcome: Mean Score on the Beck Depression Inventory (BDI) at the End of the Active and Placebo Periods
Description: The Beck Depression Inventory (BDI) is a 21-item test presented in multiple-choice format, which measures presence and degree of depression in adolescents and adults. The BDI evaluates 21 symptoms of depression. The 21 items cover sadness, pessimism, past failure, self-dislike, self-criticism, suicidal thoughts or wishes, crying, agitation, loss of interest, indecisiveness, worthlessness, loss of energy, changes in sleeping patterns, irritability, changes in appetite, difficulty concentrating, tiredness or fatigue, and loss of interest in sex. Each answer is scored on a scale value of 0-3 with 0 indicating absence of symptom and a 3 indicating severe symptom. The total range of possible scores is 0-63. A total score of <10 indicates no or minimal depression,10-18 indicates mild-to-moderate depression,19-29 indicates moderate-to-severe depression, and 30+ indicates severe depression.
Time Frame: Three months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 5 | 5
score on a scale | .80 (.84) | 1.8 (2.49)

5. Secondary Outcome: Mean Score on the Cancellation Task Following 3 Months on Active Drug and 3 Months on Placebo
Description: The WAIS-IV Cancellation Subtest assesses processing speed and attention. It is a timed test with two sequential forms, A & B. Each form requires the participant to scan an array of colored shapes (e.g., triangle, circle) randomly arranged. The participant is given 45 seconds to mark (i.e. cross out) as many of the two designated geometric shapes in the total array as possible. Cancellation scores are based on the number of correct responses minus the number of incorrect responses completed in the allotted time. The total correct for the two forms is converted to a single scaled score based on age-corrected normative data with a mean of 10 +/- 3 and a range of 1 to 19. The mean is 10 +/-3; thus a typical age corrected score is between 8 and 11; the higher the number the better the score. A low score (<8) is progressively more impaired, the lower the score. A high score (>12) indicates more efficiency and better attention than compared to others the same age.
Time Frame: Three months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 5 | 5
score on a scale | 7.6 (1.67) | 9.8 (.84)

6. Secondary Outcome: Mean Score on the Trail Making Test-A (TMT-A) Following 3 Months on Active Drug and 3 Months on Placebo
Description: The Trail Making Test-A (TMT-A) measures visual scanning and rote memory. The participant is asked to draw a line between 24 consecutive numbered circles randomly arranged on a page. The TMT-A is scored by how long it takes to complete the test. An average score for TMT-A is 29 seconds and a deficient score is >78 seconds.
Time Frame: Three months
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 5 | 5
Seconds | 47 (4.36) | 43.8 (12.87)

7. Secondary Outcome: Mean Score on the Trail Making Test-B (TMT-B) Following 3 Months on Active Drug and 3 Months on Placebo
Description: The Trail Making Test-B (TMT-B) measures visual scanning and executive functioning. The participant is asked to draw a line between 24 consecutive numbered and lettered circles randomly arranged on a page. The participant is required to switch between numbers and letters in consecutive order. The TMT-B is scored by how long it takes to complete the test. An average score for TMT-B is 75 seconds and a deficient score is >273 seconds.
Time Frame: Three months
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 5 | 5
Seconds | 43.4 (9.74) | 46 (4.36)

ADVERSE EVENTS:
Time Frame: Intervention 1 was 3 months, followed by a two week titration and 2 week Washout period. Intervention 2 was 3 months, followed by a two week titration and 1 day washout period.
Groups:
- Buspirone: Events occurring while participants on Buspirone x3 months
- Washout Period Following Buspirone: Events occurring during the washout period following 3 months of Buspirone
- Placebo: Events occurring while participants were taking Placebo x3 months
- Washout Period Following Placebo: Events occurring during the washout period following 3 months of Placebo
Arm/Group | Buspirone | Washout Period Following Buspirone | Placebo | Washout Period Following Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 6/7 | 4/7 | 3/5 | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buspirone (N=7) | Washout Period Following Buspirone (N=7) | Placebo (N=5) | Washout Period Following Placebo (N=5)
Confusion (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea with/without vomitting (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sleepy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (3) | 1 (1) | 1 (3) | 1 (1)
Fatigue (General disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Poor Memory (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall with seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Labile (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Chest pain (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (6) | 1 (1) | 1 (1) | 0 (0)
Lightheaded (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Poor balance (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin burn (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Combative (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Itchy eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vivid dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes